CLINICAL TRIAL: NCT00873366
Title: ¹³C - Dextromethorphan (DM) Breath Test for Determination of CYP2D6 Enzyme Activity in Patients Receiving Tamoxifen
Brief Title: Breath Test for Women Receiving Tamoxifen in the Prevention or Treatment of Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Funding issues
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC083C; P30CA015083 (NIH); MC083C (Other: Mayo Clinic Cancer Center); 08-007073 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dextromethorphan; Tamoxifen; Chromatography, High Pressure Liquid; Pharmacogenomic Testing; Optical Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dextromethorphan hydrobromide
Drug: tamoxifen citrate
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Other: pharmacological study
Procedure: fluorescence imaging

SUMMARY:
RATIONALE: A breath test that measures enzymes may be effective in identifying women in whom tamoxifen may not be effective.

PURPOSE: This clinical trial is studying a breath test to see how well it works in women receiving tamoxifen for the prevention or treatment of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the operating characteristics of the ¹³C-dextromethorphan (^13 C-DM) breath test in identifying women with breast cancer (or at high risk) who are CYP2D6-genotypic poor metabolizers.
* To examine the correlation between CYP2D6 enzyme activity (as measured by the breath test) and plasma endoxifen (and 4-hydroxyTAM) levels in patients who carry one or more CYP2D6 functional alleles.
* To examine the change in CYP2D6 enzyme activity (as measured by the ¹³C-DM breath test), in patients who start a CYP2D6 inhibitor while taking tamoxifen.
* To determine whether CYP2D6 enzyme activity (as measured by the breath test) changes over time (either as a consequence of drug-induced inhibition or other).
* To measure genetic variation in additional genes that are later identified to affect the metabolism, uptake, or distribution of tamoxifen (e.g., SULT1A1, UGT).

OUTLINE: Patients receive tamoxifen citrate for 6 months. ^13C-dextromethorphan breath tests are conducted at baseline and periodically during the 6 months.

13C-dextromethorphan breath test: Patients receive oral Alka-Seltzer® Gold (ASG; citric acid, potassium bicarbonate, and sodium bicarbonate) in water, then, 15 minutes later, another ASG dose and oral ¹³C-dextromethorphan. Patients breathe into a bag 1-2 times, and the is bag sealed. ¹³CO_2 levels in the bags are measured.

Blood samples are collected at baseline and periodically for pharmacogenetic and pharmacokinetic studies by reverse phase HPLC with fluorescence detection.

After completion of study therapy, patients are followed annually for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Eligible to receive tamoxifen for 6 months for either the prevention or treatment of non-invasive or invasive, stage I-III breast cancer
* CYP2D6 genotype known

  * Patients determined to be CYP2D6 poor metabolizers (by determination of a genotype test by their Mayo physician prior to study registration) are eligible to proceed with the initial breath test only
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy > 6 months
* No known impaired hepatic activity defined as ≥ grade 3 AST, alkaline phosphatase, or total bilirubin
* No pulmonary disease (e.g., asthma or other respiratory disease) associated with hypercapnia
* No uncontrolled metabolic disease (e.g., diabetes in the presence of gastroparesis, uncontrolled congestive heart failure, or uncontrolled gastrointestinal disorders [e.g., GERD])
* No prior adverse reaction to dextromethorphan
* No history of chronic liver disease (e.g., hepatitis B or hepatitis C, alcoholic liver disease, cirrhosis, or fibrotic disease)
* Able and willing to fast overnight prior to the study session
* Willing to return to Mayo Clinic for follow-up
* Willing to provide biologic specimens

PRIOR CONCURRENT THERAPY:

* More than 24 hours since prior medications known to slow gastric emptying or gastrointestinal motility (e.g., alcohol, opioid analgesics, anticholinergics [e.g., antihistamines], and loperamide)
* More than 4 weeks since prior and no concurrent CYP2D6 inhibitors or concurrent serotonin-reuptake inhibitors known to be potent CYP2D6 inhibitors (e.g.,paroxetine [Paxil®] and fluoxetine [Prozac®]

  * If mild to moderate inhibitors of CYP2D6 are medically necessary, patients may go back on after the 8-week time point
* More than 4 weeks since prior and no concurrent monoamine-oxidase inhibitors (e.g., furazolidone, phenelzine, procarbazine, selegiline, and tranylcypromine)

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Female breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-05; Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, M.D., Study Chair — Mayo Clinic; Donald W. Northfelt, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety one women and one man were enrolled between May 2009 and September 2011.
Pre-assignment Details: Six women withdrew consent prior to the start of testing. Another 9 participants were excluded from the analysis cohort due to: non-adherence to tamoxifen (N=2), use of a CYP2D6 inhibitor (N=1) and lack of sufficient samples for ¹³Cdextromethorphan analysis (N=6).
Groups:
- ¹³C-DM-BT: Participants who have provided blood samples and underwent a ¹³Cdextromethorphan breath test (¹³C-DM-BT) on day 1, once during week 8-10 following initiation of tamoxifen, and once during either month 5-6 post tamoxifen initiation.
Period: Overall Study
Arm/Group | ¹³C-DM-BT
Started | 77
Completed | 71
Not Completed | 6
Not completed — Off tamoxifen for reconstructive surgery | 1
Not completed — Off tamoxifen due to side effects | 2
Not completed — Refused to continue DM-BT testing | 3

BASELINE CHARACTERISTICS:
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 77
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 86]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 74
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 73
  1=Symptomatic and fully ambulatory | 4
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 26.8 [18.9 to 47.8]
Disease Status [Count of Participants; unit: Participants]
  Noninvasive Breast Cancer (DCIS) | 4
  Invasive Breast Cancer in Adjuvant | 72
  Invasive Breast Cancer in Metastatic | 1

OUTCOME MEASURES:

1. Primary Outcome: Operating Characteristics of the ¹³C-dextromethorphan (13C-DM) Breath Test in Identifying Those Who Are CYP2D6 Genotypic Poor Metabolizers
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The distribution of CYP2D6 genotypes grouped by CYP2D6 metabolism phenotype for each participants are summarized below.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 77
Participants
  EM/UM (*1/*2AXN) | 1
  EM/UM (*1/*1XN) | 1
  IM/UM (*41/*2AXN) | 1
  EM/EM (*1/*1) | 12
  EM/EM (*1/*2A) | 13
  EM/EM (*1/*2) | 2
  EM/EM (*2/*2) | 1
  EM/EM (*2A/*2A) | 2
  EM/IM (*1/*9) | 2
  EM/IM (*1/*10) | 3
  EM/IM (*1/*41) | 7
  EM/IM (*2A/*9) | 1
  EM/IM (*2A/*41) | 2
  EM/PM (*1/*3) | 1
  EM/PM (*1/*4) | 8
  EM/PM (*2/*4) | 1
  EM/PM (*2/*4XN) | 1
  EM/PM (*2A/*4) | 6
  EM/PM (*2A/*5) | 1
  EM/PM (*2A/*6) | 1
  IM/IM (*41/*41) | 1
  IM/PM (*3/*41) | 1
  IM/PM (*4/*9) | 1
  IM/PM (*4/*10) | 1
  IM/PM (*4/*41) | 4
  PM/PM (*3/*4) | 1
  PM/PM (*4/*4) | 1

2. Secondary Outcome: Spearman's Rank Correlation Coefficient Between CYP2D6 Genotype and ¹³Cdextromethorphan Breath Test (DM-BT)
Description: Spearman rank order correlation coefficients were used to assess the strength of the association between CYP2D6 genotype activity score and DM-BT values.
Time Frame: Baseline, 3 month and 6 month
Population: All eligible participants with DM-BT values.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 77
Correlation coefficient
  Baseline | 0.55
  3 Month: number analyzed (Participants) | 60
  3 Month | 0.58
  6 Month: number analyzed (Participants) | 55
  6 Month | 0.55

3. Secondary Outcome: Spearman's Rank Correlation Coefficient Between CYP2D6 Activity Score and Endoxifen Steady State Concentrations (Endx Css)
Description: Spearman rank order correlation coefficients were used to assess the strength of the association between CYP2D6 genotype activity score and Endx Css
Time Frame: 3 Month and 6 Month
Population: All eligible participants with Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
Correlation coefficient
  3 Month | 0.47
  6 Month: number analyzed (Participants) | 54
  6 Month | 0.56

4. Secondary Outcome: Spearman's Rank Correlation Coefficient Between CYP2D6 Activity Score and Endoxifen/N-desmethyl-tamoxifen (Endx/NDMT) Ratio
Description: Spearman rank order correlation coefficients were used to assess the strength of the association between CYP2D6 genotype activity score and Endx/NDMT ratio
Time Frame: 3 Month and 6 Month
Population: All eligible participants with Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
Correlation coefficient
  3 Month | 0.60
  6 Month: number analyzed (Participants) | 54
  6 Month | 0.61

5. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Baseline DM-BT and 3 Month Endoxifen Steady State Concentrations
Description: Spearman rank order correlation coefficients were used to assess the strength of the association between baseline ¹³Cdextromethorphan breath test (DM-BT) and Endoxifen steady state concentrations (Endx Css)
Time Frame: Baseline, 3 month
Population: All eligible participants with DM-BT values and Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
Correlation coefficient | 0.6

6. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Baseline DM-BT and 3 Month Endoxifen/N-desmethyl-tamoxifen (Endx/NDMT) Ratio
Description: Spearman rank order correlation coefficients were used to assess the strength of the association between baseline ¹³Cdextromethorphan breath test (DM-BT) and Endoxifen/N-desmethyl-tamoxifen (Endx/NDMT) Ratio
Time Frame: Baseline, 3 month
Population: All eligible participants with DM-BT values and Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
Correlation coefficient | 0.56

7. Secondary Outcome: Spearman's Rank Correlation Coefficient Between 3 Month DM-BT and 3 Month Endoxifen Steady State Concentrations
Description: as for outcome 5
Time Frame: 3 month
Population: All eligible participants with DM-BT values and Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 56
Correlation coefficient | 0.51

8. Secondary Outcome: Spearman's Rank Correlation Coefficient Between 6 Month DM-BT and 6 Month Endoxifen Steady State Concentrations
Description: as for outcome 5
Time Frame: 6 month
Population: All eligible participants with DM-BT values and Endoxifen pharmacokinetics data.
Measure: Number; unit: Correlation coefficient
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 53
Correlation coefficient | 0.54

9. Secondary Outcome: Median of 3 Month Tamoxifen Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 3 month Tamoxifen steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 3 Month
Population: All eligible participants with pharmacokinetic data available. Data was not collected for the one participant with CYP2D6 phenotype group as IM/UM.
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 219.6 [111.3 to 327.9]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 233.8 [114.8 to 275.0]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 272.3 [NA to NA] — Only one participant has the data.
  PM/EM: number analyzed (Participants) | 16
  PM/EM | 257.7 [163.0 to 514.1]
  EM/IM: number analyzed (Participants) | 10
  EM/IM | 279.1 [135.8 to 416.5]
  EM/EM: number analyzed (Participants) | 22
  EM/EM | 201.0 [134.7 to 401.4]
  IM/UM: number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 1
  EM/UM | 313.3 [NA to NA] — Only one participant has the data.

10. Secondary Outcome: Median of 6 Month Tamoxifen Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 6 month Tamoxifen steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 6 Month
Population: as for outcome 9
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 54
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 194.0 [149.3 to 238.7]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 200.5 [117.3 to 295.6]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 279.2 [NA to NA] — There is only one participant with the data.
  PM/EM: number analyzed (Participants) | 15
  PM/EM | 259.7 [47.2 to 436.6]
  EM/IM: number analyzed (Participants) | 8
  EM/IM | 234.7 [128.7 to 318.6]
  EM/EM: number analyzed (Participants) | 21
  EM/EM | 179.7 [96.6 to 460.5]
  IM/UM: number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 2
  EM/UM | 301.4 [260.7 to 342.1]

11. Secondary Outcome: Median of 3 Month N-desmethyl-tamoxifen (NDMT) Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 3 month NDMT steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 3 Month
Population: as for outcome 9
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 633.3 [429.0 to 837.7]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 578.0 [387.6 to 786.2]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 691.6 [NA to NA] — There is only one participant with the data.
  PM/EM: number analyzed (Participants) | 16
  PM/EM | 643.0 [514.6 to 885.1]
  EM/IM: number analyzed (Participants) | 10
  EM/IM | 630.7 [362.5 to 899.8]
  EM/EM: number analyzed (Participants) | 22
  EM/EM | 457.8 [325.4 to 766.7]
  IM/Ultrarapid Metabolism (UM): number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 1
  EM/UM | 576.9 [NA to NA] — There is only one participant with the data.

12. Secondary Outcome: Median of 6 Month N-desmethyl-tamoxifen (NDMT) Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 6 month NDMT steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 6 Month
Population: All eligible participants with Endoxifen pharmacokinetics data. Data was not collected for the one participant with CYP2D6 phenotype group as IM/UM.
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 54
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 554.6 [438.5 to 670.7]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 542.4 [296.2 to 813.6]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 718.2 [NA to NA] — There is only one participant with the data.
  PM/EM: number analyzed (Participants) | 15
  PM/EM | 546.5 [232.7 to 979.5]
  EM/IM: number analyzed (Participants) | 8
  EM/IM | 525.9 [373.2 to 913.8]
  EM/EM: number analyzed (Participants) | 21
  EM/EM | 401.8 [280.9 to 867.7]
  IM/UM: number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 2
  EM/UM | 552.9 [481.2 to 624.5]

13. Secondary Outcome: Median of 3 Month 4-hydroxy-tamoxifen (4HT) Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 3 month 4HT steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 3 Month
Population: All eligible participants with pharmacokinetics data. Data was not collected for the one participant with CYP2D6 phenotype group as IM/UM.
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 3.13 [2.79 to 3.47]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 1.5 [1.1 to 3.45]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 3.52 [NA to NA] — There is only one participant with the data.
  PM/EM: number analyzed (Participants) | 16
  PM/EM | 3.62 [2.08 to 8.77]
  EM/IM: number analyzed (Participants) | 9
  EM/IM | 5.41 [2.75 to 16.82]
  EM/EM: number analyzed (Participants) | 23
  EM/EM | 3.64 [1.38 to 20.05]
  IM/UM: number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 1
  EM/UM | 4.21 [NA to NA] — There is only one participant with the data.

14. Secondary Outcome: Median of 6 Month 4-hydroxy-tamoxifen (4HT) Steady State Plasma Concentrations According to CYP2D6 Phenotype Group
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 6 month 4HT steady state plasma concentrations for each CYP2D6 phenotype group are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 6 Month
Population: as for outcome 9
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 54
nM
  PM/PM: number analyzed (Participants) | 2
  PM/PM | 3.17 [2.15 to 4.19]
  IM/PM: number analyzed (Participants) | 5
  IM/PM | 1.69 [1.37 to 3.02]
  IM/IM: number analyzed (Participants) | 1
  IM/IM | 1.5 [NA to NA] — There is only one participant with the data.
  PM/EM: number analyzed (Participants) | 15
  PM/EM | 3.81 [1.37 to 12.07]
  EM/IM: number analyzed (Participants) | 8
  EM/IM | 5.86 [2.48 to 14.10]
  EM/EM: number analyzed (Participants) | 21
  EM/EM | 2.96 [1.18 to 14.1]
  IM/UM: number analyzed (Participants) | 0
  EM/UM: number analyzed (Participants) | 2
  EM/UM | 5.38 [5.24 to 5.51]

15. Secondary Outcome: Median of 3 Month Endoxifen Steady State Concentrations (Endx Css) According to CYP2D6 Phenotype Group and Activity Score
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 3 month Endx Css for each CYP2D6 phenotype group and the corresponding activity score are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 3 Month
Population: as for outcome 12
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 57
nM
  EM/UM (3.0): number analyzed (Participants) | 1
  EM/UM (3.0) | 23.6 [NA to NA] — There is only one participant with the data.
  IM/UM (2.5): number analyzed (Participants) | 0
  EM/EM (2.0): number analyzed (Participants) | 22
  EM/EM (2.0) | 30.5 [9.1 to 74.3]
  EM/IM (1.5): number analyzed (Participants) | 10
  EM/IM (1.5) | 27.9 [17.0 to 44.7]
  IM/IM (1.0): number analyzed (Participants) | 1
  IM/IM (1.0) | 11.5 [NA to NA] — There is only one participant with the data.
  EM/PM (1.0): number analyzed (Participants) | 16
  EM/PM (1.0) | 21.5 [8.6 to 50.9]
  IM/PM (0.5): number analyzed (Participants) | 5
  IM/PM (0.5) | 6.1 [4.3 to 8.5]
  PM/PM (0): number analyzed (Participants) | 2
  PM/PM (0) | 5.5 [4.6 to 6.4]

16. Secondary Outcome: Median of 6 Month Endoxifen Steady State Concentrations (Endx Css) According to CYP2D6 Phenotype Group and Activity Score
Description: Participants were classified as having CYP2D6 decreased or non-decreased metabolism based on genotype and the co-prescription of inhibitors of the enzyme system.
  The specific phenotype, alleles and their associated activity score (AS) assessed were as follows:
  Ultrarapid metabolism (UM) or AS=2.0 (*1XN or *2XN), Extensive metabolism (EM) or AS=1.0 (*1, *2, and *2A), Intermediate metabolism (IM) or AS=0.5 (*9, *10, *17 and *41), and Poor metabolism (PM) or AS=0.0 (3, *4, *5, *7, *8, *11, and *12). The median of 6 month Endx Css for each CYP2D6 phenotype group and the corresponding activity score are summarized below. Refer to Outcome Measure 1 Data Table for details on the combination of genotype for each participant that are defined for each CYP2D6 phenotype group.
Time Frame: 6 Month
Population: as for outcome 12
Measure: Median (Full Range); unit: nM
Arm/Group | ¹³C-DM-BT
Number analyzed (Participants) | 54
nM
  EM/UM (3.0): number analyzed (Participants) | 2
  EM/UM (3.0) | 38.5 [23.1 to 53.9]
  IM/UM (2.5): number analyzed (Participants) | 0
  EM/EM (2.0): number analyzed (Participants) | 21
  EM/EM (2.0) | 26.7 [10.9 to 72.9]
  EM/IM (1.5): number analyzed (Participants) | 8
  EM/IM (1.5) | 30.4 [16.1 to 38.3]
  IM/IM (1.0): number analyzed (Participants) | 1
  IM/IM (1.0) | 11.3 [NA to NA] — There is only one participant with the data.
  EM/PM (1.0): number analyzed (Participants) | 15
  EM/PM (1.0) | 19.1 [4.8 to 53.2]
  IM/PM (0.5): number analyzed (Participants) | 5
  IM/PM (0.5) | 4.7 [2.9 to 12.0]
  PM/PM (0): number analyzed (Participants) | 2
  PM/PM (0) | 6.7 [6.4 to 7.1]

ADVERSE EVENTS:
Time Frame: 6 month
Description: All eligible participants with adverse events data reported. Adverse events data were not available on 7 participants.
Arm/Group | ¹³C-DM-BT
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ¹³C-DM-BT (N=70)
Dizziness (Nervous system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes